CLINICAL TRIAL: NCT01029704
Title: A Phase II, Four-week, Multi-center, Double-blind, Placebo-controlled Parallel Group Study to Evaluate the Safety and Efficacy of EGT0001442 in Subjects With Type 2 Diabetes Mellitus With an Ascending Dose Safety and Pharmacokinetic Evaluation Period
Brief Title: Safety and Efficacy Study of EGT0001442 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THR-1442-C-402
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGT0001442 (Experimental)
  Interventions: Drug: EGT0001442
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo capsules to match EGT0001442

INTERVENTIONS:
Drug: EGT0001442 — Segment 1 is a single center, open labeled, ascending dose study in diabetic subjects who will receive 5, 10, 20, or 50 mg of EGT0001442 capsules orally once daily for 28 days.
  Segment 2 is a multi-center, double-blind, placebo-controlled parallel group study. Diabetic subjects will be randomly assigned to receive oral EGT0001442 at 5, 10, 20, or 50 mg/day for 28 days.
  Other Names: Human SGLT2 inhibitor
  Arms: EGT0001442
Drug: Placebo capsules to match EGT0001442 — Segment 1: Not applicable.
  Segment 2: Diabetic subjects will be randomly assigned to receive oral placebo once daily for 28 days.
  Other Names: Human SGLT2 inhibitor
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the effect of EGT0001442 on fasting plasma glucose after 28 days of treatment in subjects with type 2 diabetes.

The study also assessed the pharmacokinetics, safety and tolerability of EGT0001442, the effect on weight and HbA1c as well as the effect EGT0001442 has on the amount of glucose produced in the body by the urine.

DETAILED DESCRIPTION:
This was a phase 2 study to evaluate the efficacy of

EGT0001442. The study included two segments:

Segment 1 was a single center, open labeled, ascending dose study in 4 groups of 5 diabetic subjects per group who received 5, 10, 20, or 50 mg of EGT0001442 capsules orally once daily for 28 days. The subjects were in clinic for the first 3 days for safety and PK evaluation.

Segment 2 was a multi-center, double-blind, placebo-controlled parallel group study. One hundred and thirty one subjects in 5 parallel groups of approximately 25 diabetic subjects per group were randomly assigned to receive oral EGT0001442 at 5, 10, 20, or 50 mg/day or placebo once daily for 28 days in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 70 years diagnosed with type 2 diabetes.
* Body mass index (BMI) between 18 kg/m2 and 37 kg/m2 (inclusive).
* HbA1c levels between 6.5 and 9.5 (inclusive) where the upper limit of normal for the HbA1c assay is 6.4% or HbA1c levels between 6.2 and 9.5% (inclusive) where the upper limit of normal for the HbA1c assay is 6.1%.
* Fasting plasma glucose levels between 126 and 270 mg/dL (7 - 15 mmol/L, inclusive) while on diabetic medications.
* Treatment naïve subjects with HbA1c between 6.5 and 9.5 and fasting plasma glucose between 126 and 270 mg/dL (7 - 15 mmol/L).
* If taking drugs for diabetes, must be medically able and willing to discontinue diabetic medications for the duration of the study.
* Female subjects must be surgically sterilized or postmenopausal.

Exclusion Criteria:

* Type 1 diabetes or diabetes treated with insulin injection.
* Insulin therapy or oral antidiabetic medication other than metformin, sitagliptin, saxagliptin, a sulfonylurea or combination of these.
* Sitting blood pressure above 150/95 mmHg on two evaluations at least 10 minutes apart at screening.
* Positive results on screen for drugs of abuse.
* Previous treatment with an investigational drug within 30 days or 7 half-lives, whichever is longer.
* Previous treatment with EGT0001474 or EGT0001442.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason W Freeman, M.D., Study Chair — Massachusetts General Hospital
Locations (12):
- United States (9):
  - Research Site #10, Birmingham, Alabama
  - Research Site #04, National City, California
  - Research Site #12, Denver, Colorado
  - Research Site #07, Miami, Florida
  - Research Site #08, Miami, Florida
  - Research Site #06, Reading, Pennsylvania
  - Research Site #11, DeSoto, Texas
  - Research Site #01, San Antonio, Texas
  - Research Site #15, San Antonio, Texas
- Canada (3):
  - Research Site #03, Brampton, Ontario
  - Research Site #13, London, Ontario
  - Research Site #02, Mississauga, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Segment 1 (Dose Escalation): EGT0001442 5mg; Segment 2 (Double-blind): EGT0001442 5mg: Received 5mg of EGT0001442 once daily for 28 days
- Segment 1 (Dose Escalation): EGT0001442 10mg; Segment 2 (Double-blind): EGT0001442 10mg: Received 10mg of EGT0001442 once daily for 28 days
- Segment 1 (Dose Escalation): EGT0001442 20mg; Segment 2 (Double-blind): EGT0001442 20mg: Received 20mg of EGT0001442 once daily for 28 days
- Segment 1 (Dose Escalation): EGT0001442 50mg; Segment 2 (Double-blind): EGT0001442 50mg: Received 50mg of EGT0001442 once daily for 28 days
- Segment 2 (Double-blind): Placebo: Received placebo once daily for 28 days
Period: Overall Study
Arm/Group | Segment 1 (Dose Escalation): EGT0001442 5mg | Segment 1 (Dose Escalation): EGT0001442 10mg | Segment 1 (Dose Escalation): EGT0001442 20mg | Segment 1 (Dose Escalation): EGT0001442 50mg | Segment 2 (Double-blind): Placebo | Segment 2 (Double-blind): EGT0001442 5mg | Segment 2 (Double-blind): EGT0001442 10mg | Segment 2 (Double-blind): EGT0001442 20mg | Segment 2 (Double-blind): EGT0001442 50mg
Started | 5 | 5 | 5 | 5 | 28 | 24 | 23 | 28 | 26
Completed | 5 | 5 | 5 | 5 | 23 | 20 | 19 | 22 | 25
Not Completed | 0 | 0 | 0 | 0 | 5 | 4 | 4 | 6 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 2 | 0
Not completed — Withdrawn due to major protocol violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Segment 1 (Dose Escalation): EGT0001442 5mg | Segment 1 (Dose Escalation): EGT0001442 10mg | Segment 1 (Dose Escalation): EGT0001442 20mg | Segment 1 (Dose Escalation): EGT0001442 50mg | Segment 2 (Double-blind): Placebo | Segment 2 (Double-blind): EGT0001442 5mg | Segment 2 (Double-blind): EGT0001442 10mg | Segment 2 (Double-blind): EGT0001442 20mg | Segment 2 (Double-blind): EGT0001442 50mg | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 28 | 24 | 23 | 28 | 26 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Segment 1 only applies to Dose Escalation group. Segment 2 only applies to Double-blind treatment group.
  years
    Segment 1: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 20
    Segment 1 | 62.2 (7.9) | 49.4 (14.2) | 51.4 (11.7) | 53.2 (5.8) |  |  |  |  |  | 54.1 (10.8)
    Segment 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 24 | 23 | 28 | 26 | 129
    Segment 2 |  |  |  |  | 58.7 (7.3) | 57.8 (6.9) | 54.9 (9) | 59 (7.1) | 54.7 (6.7) | 57.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Segment 1 only applies to Dose Escalation group. Segment 2 only applies to Double-blind treatment group.
  Participants
    Segment 1: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 20
    Segment 1: Female | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 6
    Segment 1: Male | 4 | 4 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 14
    Segment 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 24 | 23 | 28 | 26 | 129
    Segment 2: Female |  |  |  |  | 11 | 9 | 12 | 12 | 18 | 62
    Segment 2: Male |  |  |  |  | 17 | 15 | 11 | 16 | 8 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Segment 1 only applies to Dose Escalation group. Segment 2 only applies to Double-blind treatment group.
  Participants
    Segment 1: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 20
    Segment 1: Hispanic or Latino | 4 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 15
    Segment 1: Not Hispanic or Latino | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 5
    Segment 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Segment 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 24 | 23 | 28 | 26 | 129
    Segment 2: Hispanic or Latino |  |  |  |  | 20 | 16 | 15 | 19 | 19 | 89
    Segment 2: Not Hispanic or Latino |  |  |  |  | 8 | 8 | 8 | 9 | 7 | 40
    Segment 2: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Segment 1 only applies to Dose Escalation group. Segment 2 only applies to Double-blind treatment group.
  Participants
    Segment 1: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 20
    Segment 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Segment 1: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Segment 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Segment 1: Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
    Segment 1: White | 5 | 5 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 18
    Segment 1: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Segment 1: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Segment 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 24 | 23 | 28 | 26 | 129
    Segment 2: American Indian or Alaska Native |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
    Segment 2: Asian |  |  |  |  | 5 | 2 | 3 | 4 | 1 | 15
    Segment 2: Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
    Segment 2: Black or African American |  |  |  |  | 2 | 2 | 1 | 1 | 0 | 6
    Segment 2: White |  |  |  |  | 21 | 20 | 19 | 22 | 24 | 106
    Segment 2: More than one race |  |  |  |  | 0 | 0 | 0 | 1 | 1 | 2
    Segment 2: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] — Population: Segment 1 only applies to Dose Escalation group. Segment 2 only applies to Double-blind treatment group.
  cm
    Segment 1: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 20
    Segment 1 | 172.04 (11.49) | 167.34 (11.42) | 163.74 (9.10) | 172.80 (9.00) |  |  |  |  |  | 168.98 (10.20)
    Segment 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 24 | 23 | 28 | 26 | 129
    Segment 2 |  |  |  |  | 167.76 (11.09) | 170.15 (9.32) | 167.50 (9.83) | 166.71 (9.60) | 164.92 (10.98) | 167.36 (10.19)
Weight [Mean (Standard Deviation); unit: kg] — Population: Segment 1 only applies to Dose Escalation group. Segment 2 only applies to Double-blind treatment group.
  kg
    Segment 1: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 20
    Segment 1 | 91.04 (14.48) | 83.72 (9.86) | 92.18 (16.65) | 87.22 (12.81) |  |  |  |  |  | 88.54 (13.01)
    Segment 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 24 | 23 | 28 | 26 | 129
    Segment 2 |  |  |  |  | 84.34 (15.83) | 86.75 (13.53) | 81.40 (15.03) | 81.03 (12.17) | 84.18 (17.61) | 83.51 (14.86)
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: Segment 1 only applies to Dose Escalation group. Segment 2 only applies to Double-blind treatment group.
  kg/m2
    Segment 1: number analyzed (Participants) | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 20
    Segment 1 | 30.58 (1.85) | 30.00 (3.39) | 34.18 (3.58) | 29.14 (2.94) |  |  |  |  |  | 30.98 (3.40)
    Segment 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 28 | 24 | 23 | 28 | 26 | 129
    Segment 2 |  |  |  |  | 29.77 (3.03) | 29.96 (3.98) | 28.91 (4.02) | 29.10 (3.30) | 30.75 (4.47) | 29.70 (3.77)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Fasting Plasma Glucose (FPG) From Baseline at Week 4 for Segment 2 of the Study
Description: Fasting glucose levels were measured at four time points; At day -2, day 1, day 27 and day 29 (24-h after the last dose). Baseline is defined as the mean of FPG values on day -2 and day 1. End of treatment is defined as the mean of FPG values on day 27 and day 29. Changes in the FPG during the study period was calculated by subtracting the Baseline FPG from End of Treatment FPG.
Time Frame: Baseline; Day -2 and Day 1. End of Treatment: Day 27 and Day 29
Population: Subjects participated in Segment 2 of the study were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Placebo: Received no drug (EGT0001442) during 28 days
- EGT0001442 5mg: Received 5mg of EGT0001442 per day for 28 days
- EGT0001442 10mg: Received 10mg of EGT0001442 per day for 28 days
- EGT0001442 20mg: Received 20mg of EGT0001442 per day for 28 days
- EGT0001442 50mg: Received 50mg of EGT0001442 per day for 28 days
Arm/Group | Placebo | EGT0001442 5mg | EGT0001442 10mg | EGT0001442 20mg | EGT0001442 50mg
Number analyzed (Participants) | 28 | 24 | 23 | 28 | 26
mg/dL | -12.595 (7.025) | -29.518 (7.767) | -30.429 (8.386) | -32.586 (7.305) | -44.605 (7.299)
Statistical Analysis 1: Comparison: Placebo vs EGT0001442 5mg; Test type: Superiority; p = 0.0989, ANCOVA — P-values are from two-sided test at 5% level; Analysis is based on ANCOVA with change from baseline as dependent variable and treatment as fixed effect and baseline and center as covariate; Difference of LS Means = -16.923, 95% CI 2-sided [-37.076 to 3.230]
Statistical Analysis 2: Comparison: Placebo vs EGT0001442 10mg; Test type: Superiority; p = 0.0964, ANCOVA — P-values are from two-sided test at 5% level; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -17.834, 95% CI 2-sided [-38.909 to 3.242]
Statistical Analysis 3: Comparison: Placebo vs EGT0001442 20mg; Test type: Superiority; p = 0.0465, ANCOVA — P-values are from two-sided test at 5% level; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -19.991, 95% CI 2-sided [-39.670 to -0.312]
Statistical Analysis 4: Comparison: Placebo vs EGT0001442 50mg; Test type: Superiority; p = 0.0015, ANCOVA — P-values are from two-sided test at 5% level; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -32.010, 95% CI 2-sided [-51.487 to -12.533]

2. Primary Outcome: Pharmacokinetics of EGT0001442 (Cmax) at 4 Dose Levels at Week 4
Description: Blood samples were collected during Segment 1 at pre-dose and at 30 minutes and 1, 2, 3, 4, 6, 8, 10, 12 and 24 h (day 2), and 48 h (day 3) post dose for the determination of EGT0001442. Plasma concentrations of EGT0001442 were measured using a validated HPLC/MS-MS method and PK parameters were calculated by standard noncompartmental methods.
Time Frame: Pre-dose to 48 h post-dose
Population: 20 subjects in Segment 1 of the study were included in the analysis. The PK study was not included in Segment 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Segment 1 (Dose Escalation): EGT0001442 5mg | Segment 1 (Dose Escalation): EGT0001442 10mg | Segment 1 (Dose Escalation): EGT0001442 20mg | Segment 1 (Dose Escalation): EGT0001442 50mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
ng/mL | 40.42 (15.21) | 83.38 (30.93) | 164.20 (40.21) | 541.20 (192.20)

3. Secondary Outcome: Change in the Body Weight From Baseline at Week 4
Description: Changes in the body weight during the study period was calculated by subtracting body weight on day 1 from body weight at the end of treatment on day 29.
Time Frame: Baseline and Day 29
Population: Subjects participated in Segment 2 of the study were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Placebo | EGT0001442 5mg | EGT0001442 10mg | EGT0001442 20mg | EGT0001442 50mg
Number analyzed (Participants) | 28 | 24 | 23 | 28 | 26
Kg | 0.258 (0.304) | -1.176 (0.345) | -0.779 (0.346) | -1.796 (0.324) | -0.914 (0.315)
Statistical Analysis 1: Comparison: Placebo vs EGT0001442 5mg; Test type: Superiority; p = 0.0025, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -1.434, 95% CI 2-sided [-2.349 to -0.520]
Statistical Analysis 2: Comparison: Placebo vs EGT0001442 10mg; Test type: Superiority; p = 0.0269, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -1.037, 95% CI 2-sided [-1.952 to -0.122]
Statistical Analysis 3: Comparison: Placebo vs EGT0001442 20mg; Test type: Superiority; p < 0.0001, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -2.054, 95% CI 2-sided [-2.938 to -1.170]
Statistical Analysis 4: Comparison: Placebo vs EGT0001442 50mg; Test type: Superiority; p = 0.0090, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -1.172, 95% CI 2-sided [-2.044 to -0.301]

4. Secondary Outcome: Changes in Hemoglobin A1c (HbA1c) From Baseline at Week 4
Description: HbA1c levels were measured at two time points; on day 1 and day 29 (end of treatment). Changes in the HbA1c level during the study period was calculated by subtracting HbA1c level on day 1 from HbA1c level at the end of treatment (day 29)
Time Frame: Baseline and Day 29
Population: Subjects participated in Segment 2 of the study were included in the analysis.
Measure: Geometric Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | EGT0001442 5mg | EGT0001442 10mg | EGT0001442 20mg | EGT0001442 50mg
Number analyzed (Participants) | 28 | 24 | 23 | 28 | 26
percentage of HbA1c | 0.178 (0.107) | -0.176 (0.122) | 0.022 (0.123) | 0.173 (0.115) | -0.167 (0.112)
Statistical Analysis 1: Comparison: Placebo vs EGT0001442 5mg; Test type: Superiority; p = 0.0281, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.353, 95% CI 2-sided [-0.668 to -0.039]
Statistical Analysis 2: Comparison: Placebo vs EGT0001442 10mg; Test type: Superiority; p = 0.3215, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.155, 95% CI 2-sided [-0.464 to 0.154]
Statistical Analysis 3: Comparison: Placebo vs EGT0001442 20mg; Test type: Superiority; p = 0.9776, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.004, 95% CI 2-sided [-0.304 to 0.295]
Statistical Analysis 4: Comparison: Placebo vs EGT0001442 50mg; Test type: Superiority; p = 0.0242, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.344, 95% CI 2-sided [-0.642 to -0.046]

5. Secondary Outcome: Change in Urinary Glucose Excretion From Baseline to Day 1 and Day 28
Description: Urinary glucose levels were measured at three time points; on Day 0 (baseline), Day 1 and Day 28 (end of treatment). Changes in the urinary glucose level during the study period was calculated by reducing the baseline urinary glucose level (Day 1) from urinary glucose level at end of treatment (Day 28) (i.e urinary glucose level on Day 28 minus urinary glucose level on Day 1).
Time Frame: Baseline, Day 1 and Day 28
Population: Only number of subjects with data available in the specific treatment group is included
Measure: Mean (Standard Deviation); unit: g/24h
Arm/Group | Placebo | EGT0001442 5mg | EGT0001442 10mg | EGT0001442 20mg | EGT0001442 50mg
Number analyzed (Participants) | 28 | 23 | 22 | 28 | 26
g/24h
  Change in 24 h UGE from baseline to Day 1: number analyzed (Participants) | 26 | 19 | 21 | 25 | 25
  Change in 24 h UGE from baseline to Day 1 | -3.55 (13.05) | 26.21 (11.08) | 24.17 (16.89) | 25.13 (12.72) | 29.61 (20.00)
  Change in 24 h UGE from baseline to Day 28 | -0.20 (14.98) | 22.57 (16.56) | 18.71 (20.46) | 21.01 (16.43) | 26.80 (19.36)

6. Secondary Outcome: Change in FPG Following Cessation of Treatment
Description: The mean change in FPG following cessation of treatment was obtained by calculating the difference between FPG values obtained on End of treatment (average of FPG values on days 27 and 29) and on Post Treatment (average of FPG values on days 41 and 43).
Time Frame: Days 27/29 to Days 41/43
Population: Subjects participated in Segment 2 of the study and had fasting plasma glucose (FPG) values at the end of treatment (mean FPG value on days 27 and 29) and at post-treatment (mean FPG values on days 41 and 43) are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | EGT0001442 5mg | EGT0001442 10mg | EGT0001442 20mg | EGT0001442 50mg
Number analyzed (Participants) | 26 | 21 | 19 | 21 | 25
mg/dL | 0.058 (8.256) | 17.746 (8.896) | 17.148 (10.421) | 24.437 (7.989) | 20.807 (8.021)
Statistical Analysis 1: Comparison: Placebo vs EGT0001442 5mg; Test type: Superiority; p = 0.1613, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = 17.688, 95% CI 2-sided [-7.210 to 42.587]
Statistical Analysis 2: Comparison: Placebo vs EGT0001442 10mg; Test type: Superiority; p = 0.2079, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = 17.091, 95% CI 2-sided [-9.696 to 43.877]
Statistical Analysis 3: Comparison: Placebo vs EGT0001442 20mg; Test type: Superiority; p = 0.0410, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = 24.379, 95% CI 2-sided [1.028 to 47.731]
Statistical Analysis 4: Comparison: Placebo vs EGT0001442 50mg; Test type: Superiority; p = 0.0862, ANCOVA — P-values are from a two-sided test; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = 20.749, 95% CI 2-sided [-3.019 to 44.518]

7. Primary Outcome: Pharmacokinetics of EGT0001442 (AUC 0-t and 0-24) at 4 Dose Levels at Week 4
Description: as for outcome 2
Time Frame: Pre-dose to 48 h post-dose
Population: 20 subjects in Segment 1 of the study were included in the analysis. The PK study was not included in Segment 2.
  AUC0-24 values for two participants in 5 mg arm were not calculated.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Segment 1 (Dose Escalation): EGT0001442 5mg | Segment 1 (Dose Escalation): EGT0001442 10mg | Segment 1 (Dose Escalation): EGT0001442 20mg | Segment 1 (Dose Escalation): EGT0001442 50mg
Number analyzed (Participants) | 5 | 5 | 5 | 5
ng*h/mL
  AUC0-t | 334.02 (51.80) | 681.88 (74.66) | 1312.36 (487.28) | 3308.88 (785.59)
  AUC0-24: number analyzed (Participants) | 3 | 5 | 5 | 5
  AUC0-24 | 328.85 (56.07) | 548.15 (70.41) | 1076.39 (373.15) | 2755.68 (586.08)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day -7 (Visit 3; Washout monitor) to Day 43 (Visit 14; Termination)
Arm/Group | Segment 1 (Dose Escalation): EGT0001442 5mg | Segment 1 (Dose Escalation): EGT0001442 10mg | Segment 1 (Dose Escalation): EGT0001442 20mg | Segment 1 (Dose Escalation): EGT0001442 50mg | Placebo | EGT0001442 5mg | EGT0001442 10mg | EGT0001442 20mg | EGT0001442 50mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/28 | 0/24 | 0/23 | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/28 | 1/24 | 1/23 | 0/28 | 0/26
Other Adverse Events (participants affected / at risk) | 3/5 | 3/5 | 3/5 | 2/5 | 4/28 | 3/24 | 6/23 | 6/28 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Segment 1 (Dose Escalation): EGT0001442 5mg (N=5) | Segment 1 (Dose Escalation): EGT0001442 10mg (N=5) | Segment 1 (Dose Escalation): EGT0001442 20mg (N=5) | Segment 1 (Dose Escalation): EGT0001442 50mg (N=5) | Placebo (N=28) | EGT0001442 5mg (N=24) | EGT0001442 10mg (N=23) | EGT0001442 20mg (N=28) | EGT0001442 50mg (N=26)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Segment 1 (Dose Escalation): EGT0001442 5mg (N=5) | Segment 1 (Dose Escalation): EGT0001442 10mg (N=5) | Segment 1 (Dose Escalation): EGT0001442 20mg (N=5) | Segment 1 (Dose Escalation): EGT0001442 50mg (N=5) | Placebo (N=28) | EGT0001442 5mg (N=24) | EGT0001442 10mg (N=23) | EGT0001442 20mg (N=28) | EGT0001442 50mg (N=26)
Leucopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Balanitis candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 4 | 3
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator does not have the right to publish trial results.

DOCUMENTS (1):
  • Statistical Analysis Plan (2010-05-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT01029704/SAP_000.pdf